CLINICAL TRIAL: NCT00778102
Title: A Multicentre Randomised Phase II Study to Assess the Safety and Resectability in Patients With Initially Unresectable Liver Metastases Secondary to Colorectal Cancer Receiving First-line Treatment Either With mFOLFOX-6 Plus Bevacizumab or FOLFOXIRI Plus Bevacizumab (OLIVIA)
Brief Title: A Study of Avastin (Bevacizumab) in Combination With mFOLFOX-6 or FOLFOXIRI in Patients With Metastatic Colorectal Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO18725; 2007-007863-26
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Results first posted 2015-08-07 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Irinotecan; Leucovorin; Oxaliplatin; Bevacizumab

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: 5-FU; Drug: Leucovorin; Drug: Oxaliplatin; Drug: bevacizumab [Avastin]
- 2 (Active Comparator)
  Interventions: Drug: 5-FU; Drug: Irinotecan; Drug: Leucovorin; Drug: Oxaliplatin; Drug: bevacizumab [Avastin]

INTERVENTIONS:
Drug: 5-FU — Bolus 400mg/m2, day 1 every 2 weeks
  Arms: 1
Drug: 5-FU — 3200mg/m2 46-hour continuous iv infusion, day 1 every 2 weeks
  Arms: 2
Drug: 5-FU — 2400mg/m2 46-hour continuous iv infusion, day 1 every 2 weeks
  Arms: 1
Drug: Irinotecan — 165mg/m2 1-hour iv infusion, day 1 every 2 weeks
  Arms: 2
Drug: Leucovorin — 400mg/m2 2-hour iv infusion, day 1 every 2 weeks
  Arms: 1
Drug: Leucovorin — 200mg/m2 2-hour iv infusion, day 1 every 2 weeks
  Arms: 2
Drug: Oxaliplatin — 85mg/m2 2-hour iv infusion, day 1 every 2 weeks
Drug: bevacizumab [Avastin] — 5mg/kg iv day 1 every 2 weeks

SUMMARY:
This 2 arm study will compare the resection rate of liver metastases and safety of surgery in patients with metastatic colorectal cancer and primarily unresectable liver metastases receiving treatment with Avastin in combination with 5-FU, leucovorin and oxaliplatin with irinotecan (FOLFOXIRI) or without irinotecan (mFOLFOX-6) as first line treatment. Patients will be randomized to receive Avastin (5mg/kg iv every 2 weeks) in combination with each of these two standard neoadjuvant chemotherapy regimens. The anticipated time on study treatment is until surgery, disease progression, unacceptable toxicity or patient refusal, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* unresectable liver metastasis secondary to cancer of colon or rectum;
* scheduled for standard first line chemotherapy;
* ECOG performance score of 0 or 1;
* condition feasible for major abdominal surgery after first line treatment.

Exclusion Criteria:

* diagnosis of metastatic disease >3 months prior to study entry;
* evidence of extrahepatic disease, diffuse peritoneal carcinosis or involvement of celiac lymph nodes;
* prior systemic or local treatment of metastatic disease;
* prior (neo)adjuvant chemotherapy/radiotherapy completed within 6 months prior to study entry;
* history or evidence of CNS disease unrelated to cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (18):
- Vienna, Austria
- France (7):
  - Bordeaux
  - Créteil
  - Le Mans
  - Lille
  - Lyon
  - Montpellier
  - Villejuif
- Spain (6):
  - Palma de Mallorca, Balearic Islands
  - Girona, Girona
  - Donostia / San Sebastian, Guipuzcoa
  - Santiago de Compostela, La Coruña
  - Madrid, Madrid
  - Valencia, Valencia
- United Kingdom (4):
  - London
  - Manchester
  - Metropolitan Borough of Wirral
  - Sutton

REFERENCES:
- [Derived] Cremolini C, Antoniotti C, Stein A, Bendell J, Gruenberger T, Rossini D, Masi G, Ongaro E, Hurwitz H, Falcone A, Schmoll HJ, Di Maio M. Individual Patient Data Meta-Analysis of FOLFOXIRI Plus Bevacizumab Versus Doublets Plus Bevacizumab as Initial Therapy of Unresectable Metastatic Colorectal Cancer. J Clin Oncol. 2020 Aug 20:JCO2001225. doi: 10.1200/JCO.20.01225. Online ahead of print. PMID 32816630
- [Derived] Gruenberger T, Bridgewater J, Chau I, Garcia Alfonso P, Rivoire M, Mudan S, Lasserre S, Hermann F, Waterkamp D, Adam R. Bevacizumab plus mFOLFOX-6 or FOLFOXIRI in patients with initially unresectable liver metastases from colorectal cancer: the OLIVIA multinational randomised phase II trial. Ann Oncol. 2015 Apr;26(4):702-708. doi: 10.1093/annonc/mdu580. Epub 2014 Dec 23. PMID 25538173

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab + mFOLFOX-6: Participants received a chemotherapy regimen of bevacizumab plus oxaliplatin, leucovorin, and 5-fluorouracil (5-FU) (mFOLFOX-6). Each drug was administered on Day 1 of each 2-week cycle. Dosing was as follows: bevacizumab 5 milligrams per kilogram (mg/kg) via intravenous (IV) infusion; oxaliplatin 85 milligrams per meter-squared (mg/m^2) via IV infusion; leucovorin 400 mg/m^2 via IV infusion; 5-FU 400 mg/m^2 via IV bolus; and 5-FU 2400 mg/m^2 via continuous 46-hour IV infusion. Following completion of 12 cycles, participants could discontinue oxaliplatin and continue with bevacizumab, leucovorin, and 5-FU. Treatment was continued until resectability, progressive disease (PD), unacceptable toxicity, or participant refusal.
- Bevacizumab + FOLFOXIRI: Participants received a chemotherapy regimen of bevacizumab plus oxaliplatin, irinotecan, leucovorin, and 5-FU (FOLFOXIRI). Each drug was administered on Day 1 of each 2-week cycle. Dosing was as follows: bevacizumab 5 mg/kg via IV infusion; oxaliplatin 85 mg/m^2 via IV infusion; irinotecan 165 mg/m^2 via IV infusion; leucovorin 200 mg/m^2 via IV infusion; and 5-FU 3200 mg/m^2 via continuous 46-hour IV infusion. Following completion of 12 cycles, participants were to discontinue either irinotecan, oxaliplatin, or both. Treatment was continued until resectability, PD, unacceptable toxicity, or participant refusal.
Period: Overall Study
Arm/Group | Bevacizumab + mFOLFOX-6 | Bevacizumab + FOLFOXIRI
Started | 39 | 41
Completed | 18 | 19
Not Completed | 21 | 22
Not completed — Adverse Event | 8 | 5
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Violation of Selection Criteria | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Refused Treatment | 2 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Administrative Reason | 7 | 10

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: All randomized participants. Participants were analyzed according to which treatment group they were randomized, regardless of the treatment actually received.
Groups:
- Bevacizumab + mFOLFOX-6: Participants received a chemotherapy regimen of bevacizumab plus mFOLFOX-6. Each drug was administered on Day 1 of each 2-week cycle. Dosing was as follows: bevacizumab 5 mg/kg via IV infusion; oxaliplatin 85 mg/m^2 via IV infusion; leucovorin 400 mg/m^2 via IV infusion; 5-FU 400 mg/m^2 via IV bolus; and 5-FU 2400 mg/m^2 via continuous 46-hour IV infusion. Following completion of 12 cycles, participants could discontinue oxaliplatin and continue with bevacizumab, leucovorin, and 5-FU. Treatment was continued until resectability, PD, unacceptable toxicity, or participant refusal.
- Bevacizumab + FOLFOXIRI: Participants received a chemotherapy regimen of bevacizumab plus FOLFOXIRI. Each drug was administered on Day 1 of each 2-week cycle. Dosing was as follows: bevacizumab 5 mg/kg via IV infusion; oxaliplatin 85 mg/m^2 via IV infusion; irinotecan 165 mg/m^2 via IV infusion; leucovorin 200 mg/m^2 via IV infusion; and 5-FU 3200 mg/m^2 via continuous 46-hour IV infusion. Following completion of 12 cycles, participants were to discontinue either irinotecan, oxaliplatin, or both. Treatment was continued until resectability, PD, unacceptable toxicity, or participant refusal.
- Total: Total of all reporting groups
Arm/Group | Bevacizumab + mFOLFOX-6 | Bevacizumab + FOLFOXIRI | Total
Number analyzed (Participants) | 39 | 41 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (10.32) | 61.8 (11.02) | 59.5 (10.87)
Gender [Count of Participants; unit: Participants]
  Female | 21 | 12 | 33
  Male | 18 | 29 | 47

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Resection or Residual (Microscopic or Macroscopic) Tumor
Description: Following resective surgery, participants were evaluated for complete resection (R0) or the presence of microscopic (R1) or macroscopic (R2) residual tumor. The percentage of participants within each residual tumor classification was calculated as [number of participants with R0, R1, and/or R2 divided by the total number of participants] multiplied by 100. Associated 95% confidence intervals were calculated for one-sample binomial using the Clopper-Pearson method.
Time Frame: Up to 5 years (at Screening; every 6 weeks, and within 4 weeks prior to surgery; and at time of/after surgery)
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX-6 | Bevacizumab + FOLFOXIRI
Number analyzed (Participants) | 39 | 41
percentage of participants
  R0, R1, or R2 | 48.7 [32.4 to 65.2] | 61.0 [44.5 to 75.8]
  R0 or R1 | 33.3 [19.1 to 50.2] | 51.2 [35.1 to 67.1]
  R0 | 23.1 [11.1 to 39.3] | 48.8 [32.9 to 64.9]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX-6 vs Bevacizumab + FOLFOXIRI; Difference between groups in the collective percentage of participants with R0, R1, or R2; Test type: Superiority or Other; p = 0.2707, Chi-squared; Difference in Resection Rate = 12.3, 95% CI 2-sided [-11.0 to 35.5] — Confidence interval calculated for difference based on Hauck-Anderson method

2. Secondary Outcome: Time to Resection
Description: Time to resection was defined as the time from randomization to the date of first resective surgery. For participants who did not undergo resective surgery, time to resection was censored at Day 1. Time to resection was estimated by Kaplan-Meier analysis.
Time Frame: Up to 5 years (at Screening; prior to each cycle, and within 7 days prior to surgery; and at time of surgery)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + mFOLFOX-6 | Bevacizumab + FOLFOXIRI
Number analyzed (Participants) | 39 | 41
months | 4.4 [4.1 to 5.8] | 4.3 [3.9 to 5.5]

3. Secondary Outcome: Percentage of Participants With Histopathological Response
Description: At the time of resective surgery, participants were evaluated for histopathological response as defined through pathologist review of the resected metastatic lesions, including assessment of margin status and tumor cell viability. Histopathological response classification was based upon the percentage of viable tumor cells, where 'Complete response' was considered for those with 0 percent (%) viable tumor cells, 'Major response' for those with 1% to 49% viable tumor cells, 'Minor response' for 50% to 99% viable tumor cells, and 'No response' for 100% viable tumor cells. The response could not be determined in some cases and was documented as 'Unknown.' The percentage of participants within each response category was calculated as [number of participants with a given response divided by the number of participants who completed the assessment] multiplied by 100.
Time Frame: Up to 5 years (at Screening; every 6 weeks, and within 4 weeks prior to surgery; and at time of/after surgery)
Population: ITT Population; only participants with a histopathological assessment after the first resective surgery were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX-6 | Bevacizumab + FOLFOXIRI
Number analyzed (Participants) | 14 | 21
percentage of participants
  Complete response | 0 | 4.8
  Major response | 57.1 | 47.6
  Minor response | 28.6 | 33.3
  No response | 0 | 0
  Unknown | 14.3 | 14.3

4. Secondary Outcome: Percentage of Participants With Complete or Major Histopathological Response
Description: At the time of resective surgery, participants were evaluated for histopathological response as defined through pathologist review of the resected metastatic lesions, including assessment of margin status and tumor cell viability. Histopathological response classification was based upon the percentage of viable tumor cells, as described previously. The collective percentage of participants assessed as having a complete or major response was calculated as [number of participants with complete or major response divided by the number of participants who completed the assessment] multiplied by 100. Associated 95% confidence intervals were calculated for one-sample binomial using the Clopper-Pearson method.
Time Frame: Up to 5 years (at Screening; every 6 weeks, and within 4 weeks prior to surgery; and at time of/after surgery)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX-6 | Bevacizumab + FOLFOXIRI
Number analyzed (Participants) | 14 | 21
percentage of participants | 57.1 [28.9 to 82.3] | 52.4 [29.8 to 74.3]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX-6 vs Bevacizumab + FOLFOXIRI; Difference between groups in the collective percentage of participants with complete or major histopathological response; Test type: Superiority or Other; p = 0.7817, Chi-squared; Difference in Response Rate = -4.8, 95% CI 2-sided [-43.0 to 33.5] — Confidence interval calculated for difference based on Hauck-Anderson method

5. Secondary Outcome: Percentage of Participants Experiencing Relapse Following Curative Resection
Description: Among participants with curative resection (complete resection [R0] or microscopic residual tumor [R1]), relapse was defined as the first new occurrence of cancer or death. The percentage of participants who experienced relapse was calculated as [number of participants with a relapse event divided by the number of participants initially classified as R0 or R1 following resective surgery] multiplied by 100.
Time Frame: Up to 5 years (at time of surgery; 48 hours and 4 and 12 weeks after surgery; within 4 weeks after completion of treatment; every 3 to 6 months for 1 year; then annually)
Population: ITT Population; only participants with a residual tumor classification of R0 or R1 after first resection were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX-6 | Bevacizumab + FOLFOXIRI
Number analyzed (Participants) | 13 | 21
percentage of participants | 76.9 | 57.1

6. Secondary Outcome: Relapse-Free Survival (RFS)
Description: RFS was defined as the time from curative resection (complete resection [R0] or microscopic residual tumor [R1]) to the date of first diagnosis of relapse. For participants with curative resection and without relapse, RFS was censored at the last known relapse-free assessment. RFS was estimated by Kaplan-Meier analysis.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + mFOLFOX-6 | Bevacizumab + FOLFOXIRI
Number analyzed (Participants) | 13 | 21
months | 8.1 [3.8 to 11.7] | 17.1 [12.3 to NA] — Confidence interval upper limit was not reached due to insufficient follow-up.

7. Secondary Outcome: Percentage of Participants Experiencing Death or Disease Progression
Description: PD was defined, using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0, as at least a 20% increase in the sum of the longest diameter of target lesions, or the appearance of one or more new lesions. The percentage of participants experiencing PD or death was calculated as [number of participants with event divided by the number of participants analyzed] multiplied by 100.
Time Frame: Up to 5 years (at Screening; every 6 weeks, and within 4 weeks prior to surgery; 4 and 12 weeks after surgery; and at the end of Cycles 4 and 8 if assessed as R0 or R1, or every 6 weeks until progression or resectability if assessed as R2)
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX-6 | Bevacizumab + FOLFOXIRI
Number analyzed (Participants) | 39 | 41
percentage of participants | 89.7 | 68.3

8. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined, using RECIST version 1.0, as the time from randomization to the date of first documented PD or death from any cause. PD was defined as at least a 20% increase in the sum of the longest diameter of target lesions, or the appearance of one or more new lesions. For participants without documented PD or death, PFS was censored at the time of last tumor assessment. PFS was estimated by Kaplan-Meier analysis.
Time Frame: as for outcome 7
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + mFOLFOX-6 | Bevacizumab + FOLFOXIRI
Number analyzed (Participants) | 39 | 41
months | 11.5 [9.6 to 13.6] | 18.6 [12.9 to 22.3]

9. Secondary Outcome: Percentage of Participants Who Died
Time Frame: Up to 5 years (prior to each cycle, and within 7 days prior to surgery; at time of surgery; 48 hours and 4 and 12 weeks after surgery; within 4 weeks after completion of treatment; every 3 to 6 months for 1 year; then annually)
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX-6 | Bevacizumab + FOLFOXIRI
Number analyzed (Participants) | 39 | 41
percentage of participants | 48.7 | 19.5

10. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death from any cause. For participants without an event of death, OS was censored at the last-known alive date. OS was estimated by Kaplan-Meier analysis.
Time Frame: as for outcome 9
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + mFOLFOX-6 | Bevacizumab + FOLFOXIRI
Number analyzed (Participants) | 39 | 41
months | 32.2 [21.5 to NA] — Confidence interval upper limit was not reached due to insufficient follow-up. | NA [NA to NA] — Median and corresponding confidence interval were not reached due to insufficient follow-up.

11. Secondary Outcome: Percentage of Participants With a Confirmed Best Overall Response of Complete Response (CR) or Partial Response (PR) According to RECIST Version 1.0
Description: Using RECIST version 1.0, participants were considered to have achieved CR upon the disappearance of all target and non-target lesions. Participants who achieved PR demonstrated at least a 30% decrease in the sum of the largest diameter of target lesions, taking as reference the Screening sum largest diameter. Responses were confirmed by repeat assessments no less than 4 weeks after criteria for response were first met. The collective percentage of participants with confirmed best overall response of CR or PR was calculated as [number of participants meeting RECIST criteria for CR or PR divided by the number of participants analyzed] multiplied by 100. Associated 95% confidence intervals were calculated for one-sample binomial using the Clopper-Pearson method.
Time Frame: as for outcome 7
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX-6 | Bevacizumab + FOLFOXIRI
Number analyzed (Participants) | 39 | 41
percentage of participants | 61.5 [44.6 to 76.6] | 80.5 [65.1 to 91.2]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX-6 vs Bevacizumab + FOLFOXIRI; Difference between groups in the collective percentage of participants with confirmed best overall response of CR or PR; Test type: Superiority or Other; p = 0.0612, Chi-squared; Difference in Response Rate (CR or PR) = 18.9, 95% CI 2-sided [-2.1 to 40.0] — Confidence interval calculated for difference based on Hauck-Anderson method

12. Secondary Outcome: Time to Response
Description: Time to response according to RECIST version 1.0 was defined as the time from randomization to the date of first documented CR or PR. Participants were considered to have achieved CR upon the disappearance of all target and non-target lesions. Participants who achieved PR demonstrated at least a 30% decrease in the sum of the largest diameter of target lesions, taking as reference the Screening sum largest diameter. Responses were confirmed by repeat assessments no less than 4 weeks after criteria for response were first met. For participants who did not complete a confirmatory tumor assessment, time to response was censored at the date of last tumor assessment, or if unavailable, at the date of first dose. Time to response was estimated by Kaplan-Meier analysis.
Time Frame: as for outcome 7
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + mFOLFOX-6 | Bevacizumab + FOLFOXIRI
Number analyzed (Participants) | 39 | 41
months | 3.1 [2.7 to 8.6] | 3.1 [1.9 to 3.9]

13. Secondary Outcome: Percentage of Participants With Complications Related to First Resective Surgery
Description: Complications related to the first resective surgery were evaluated using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 3.0, and classified according to severity. The NCI-CTCAE severity classification criteria are as follows: Grade 5 equals (=) resulting in death; Grade 4 = life-threatening; Grade 3 = severe; Grade 2 = moderate; and Grade 1 = mild. The percentage of participants experiencing a given adverse event (AE) by severity grade was calculated as [number of participants with an AE divided by the number of participants who underwent first resective surgery] multiplied by 100.
Time Frame: as for outcome 5
Population: Safety Population (First Surgery Subpopulation): All participants who underwent a first resective surgery and who received at least one dose of trial medication, whether prematurely withdrawn or not. Participants were analyzed according to the actual treatment they received.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX-6 | Bevacizumab + FOLFOXIRI
Number analyzed (Participants) | 19 | 25
percentage of participants
  Any complication, Total | 73.7 | 52.0
  Any complication, Grade 1 | 15.8 | 4.0
  Any complication, Grade 2 | 36.8 | 12.0
  Any complication, Grade 3 | 10.5 | 24.0
  Any complication, Grade 4 | 0 | 12.0
  Any complication, Grade 5 | 10.5 | 0
  Bleeding, Total | 15.8 | 8.0
  Bleeding, Grade 1 | 5.3 | 0
  Bleeding, Grade 2 | 5.3 | 4.0
  Bleeding, Grade 3 | 5.3 | 4.0
  Cardiovascular, Total | 10.5 | 4.0
  Cardiovascular, Grade 2 | 0 | 4.0
  Cardiovascular, Grade 3 | 5.3 | 0
  Cardiovascular, Grade 4 | 5.3 | 0
  Infections, Total | 26.3 | 32.0
  Infections, Grade 1 | 10.5 | 12.0
  Infections, Grade 2 | 5.3 | 0
  Infections, Grade 3 | 5.3 | 16.0
  Infections, Grade 4 | 5.3 | 4.0
  Liver insufficiency, Total | 10.5 | 0
  Liver insufficiency, Grade 5 | 10.5 | 0
  Neural disorder, Total | 5.3 | 0
  Neural disorder, Grade 2 | 5.3 | 0
  Noninfected perihepatic fluid collections, Total | 0 | 4.0
  Noninfected perihepatic fluid collections, Grade 2 | 0 | 4.0
  Other complication, Total | 52.6 | 28.0
  Other complication, Grade 1 | 26.3 | 8.0
  Other complication, Grade 2 | 21.1 | 8.0
  Other complication, Grade 3 | 0 | 12.0
  Other complication, Grade 4 | 5.3 | 0
  Pulmonary, Total | 5.3 | 4.0
  Pulmonary, Grade 3 | 5.3 | 4.0
  Renal impairment, Total | 10.5 | 4.0
  Renal impairment, Grade 2 | 5.3 | 4.0
  Renal impairment, Grade 4 | 5.3 | 0
  Wound healing, Total | 5.3 | 12.0
  Wound healing, Grade 1 | 5.3 | 0
  Wound healing, Grade 3 | 0 | 4.0
  Wound healing, Grade 4 | 0 | 8.0

14. Secondary Outcome: Percentage of Participants With Complications Related to Second Resective Surgery
Description: Complications related to the second resective surgery were evaluated using the NCI-CTCAE version 3.0, and classified according to severity. The NCI-CTCAE severity classification criteria are as follows: Grade 5 = resulting in death; Grade 4 = life-threatening; Grade 3 = severe; Grade 2 = moderate; and Grade 1 = mild. The percentage of participants experiencing a given AE by severity grade was calculated as [number of participants with an AE divided by the number of participants who underwent second resective surgery] multiplied by 100.
Time Frame: as for outcome 5
Population: Safety Population (Second Surgery Subpopulation): All participants who underwent a second resective surgery and who received at least one dose of trial medication, whether prematurely withdrawn or not. Participants were analyzed according to the actual treatment they received.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX-6 | Bevacizumab + FOLFOXIRI
Number analyzed (Participants) | 3 | 3
percentage of participants
  Any complication, Total | 100.0 | 66.7
  Any complication, Grade 1 | 0 | 33.3
  Any complication, Grade 2 | 66.7 | 0
  Any complication, Grade 3 | 0 | 33.3
  Any complication, Grade 3a | 33.3 | 0
  Bleeding, Total | 33.3 | 33.3
  Bleeding, Grade 1 | 0 | 33.3
  Bleeding, Grade 2 | 33.3 | 0

ADVERSE EVENTS:
Time Frame: Up to 5 years (at Screening; prior to each cycle, and within 7 days prior to surgery; at time of surgery; 48 hours and 4 and 12 weeks after surgery; within 4 weeks after completion of treatment; every 3 to 6 months for 1 year; then annually)
Description: Safety Population: All participants who received at least one dose of trial medication, whether prematurely withdrawn or not.
Arm/Group | Bevacizumab + mFOLFOX-6 | Bevacizumab + FOLFOXIRI
Serious Adverse Events (participants affected / at risk) | 24/37 | 24/40
Other Adverse Events (participants affected / at risk) | 36/37 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + mFOLFOX-6 (N=37) | Bevacizumab + FOLFOXIRI (N=40)
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 6
Ileus (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 6
Neutropenia (Blood and lymphatic system disorders) | 3 | 4
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 2
Bacterial sepsis (Infections and infestations) | 1 | 0
Campylobacter infection (Infections and infestations) | 0 | 1
Cholecystitis infective (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 2
Thrombosis (Vascular disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 2
General physical health deterioration (General disorders) | 1 | 0
Impaired healing (General disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 2 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 3
Failure to anastomose (Injury, poisoning and procedural complications) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Endoscopic retrograde cholangiopancreatography (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Pelvic fluid collection (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + mFOLFOX-6 (N=37) | Bevacizumab + FOLFOXIRI (N=40)
Diarrhoea (Gastrointestinal disorders) | 20 | 33
Nausea (Gastrointestinal disorders) | 23 | 21
Vomiting (Gastrointestinal disorders) | 14 | 25
Constipation (Gastrointestinal disorders) | 18 | 15
Abdominal pain (Gastrointestinal disorders) | 15 | 15
Dry mouth (Gastrointestinal disorders) | 7 | 8
Abdominal pain upper (Gastrointestinal disorders) | 8 | 5
Stomatitis (Gastrointestinal disorders) | 5 | 3
Toothache (Gastrointestinal disorders) | 4 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 2
Proctalgia (Gastrointestinal disorders) | 1 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 2
Flatulence (Gastrointestinal disorders) | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 22 | 19
Paraesthesia (Nervous system disorders) | 12 | 7
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 4
Headache (Nervous system disorders) | 9 | 7
Dysgeusia (Nervous system disorders) | 5 | 10
Lethargy (Nervous system disorders) | 3 | 2
Dysaesthesia (Nervous system disorders) | 3 | 2
Dizziness (Nervous system disorders) | 3 | 1
Polyneuropathy (Nervous system disorders) | 3 | 1
Asthenia (General disorders) | 14 | 16
Mucosal inflammation (General disorders) | 20 | 17
Fatigue (General disorders) | 10 | 12
Pyrexia (General disorders) | 7 | 12
Catheter site pain (General disorders) | 2 | 1
Pain (General disorders) | 1 | 2
Chest pain (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 20 | 26
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 8
Anaemia (Blood and lymphatic system disorders) | 4 | 6
Leukopenia (Blood and lymphatic system disorders) | 1 | 4
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Platelet count decreased (Investigations) | 5 | 3
Haemoglobin decreased (Investigations) | 2 | 2
White blood cell count decreased (Investigations) | 2 | 1
Gamma-glutamyltransferase increased (Investigations) | 3 | 1
Blood lactate dehydrogenase increased (Investigations) | 2 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1
Weight decreased (Investigations) | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 8 | 13
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 5 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 0
Urinary tract infection (Infections and infestations) | 4 | 4
Nasopharyngitis (Infections and infestations) | 4 | 1
Oral herpes (Infections and infestations) | 3 | 3
Rhinitis (Infections and infestations) | 1 | 2
Device related infection (Infections and infestations) | 2 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 3
Candida infection (Infections and infestations) | 2 | 0
Tracheitis (Infections and infestations) | 0 | 2
Hypertension (Vascular disorders) | 8 | 5
Hypotension (Vascular disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 7 | 2
Anxiety (Psychiatric disorders) | 2 | 1
Hypersensitivity (Immune system disorders) | 3 | 3
Vertigo (Ear and labyrinth disorders) | 2 | 2
Proteinuria (Renal and urinary disorders) | 2 | 4
Procedural pain (Injury, poisoning and procedural complications) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.